CLINICAL TRIAL: NCT00703339
Title: A Single-Dose, Dose-Escalating Study Exploring the Safety, Pharmacokinetics, and Pharmacodynamic Effects of Inhaled Treprostinil Sodium Using the Nebu-Tec OPTINEB Inhalation Device in Patients With Pulmonary Hypertension Associated With Idiopathic Pulmonary Fibrosis
Brief Title: Effects of Inhaled Treprostinil Sodium for the Treatment of Pulmonary Hypertension Associated With Idiopathic Pulmonary Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment to the trial. Very difficult population to recruit.
Sponsor: Lung Biotechnology PBC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TREINH-IPF-201
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Results first posted 2012-05-10 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2012-05

CONDITIONS: Idiopathic Pulmonary Fibrosis; Pulmonary Hypertension
Keywords: fibrosis, pulmonary; hypertension, pulmonary; exercise, aerobic
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Hypertension, Pulmonary; Pulmonary Fibrosis; Motor Activity | interventions — treprostinil; Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Treprostinil sodium for inhalation — Administration of inhaled treprostinil sodium 0.6 mg/ml in 3mL ampoules Duration of Treatment: single dose
  Dose:
  * Cohort 1: dosed at 3 breaths (18 mcg)
  * Cohort 2: dosed at 6 breaths (36 mcg)
  * Cohort 3: dosed at 9 breaths (54 mcg)
  * Cohort 4: dosed at 12 breaths (72 mcg)
  The decision to advance to the next cohort will be made after review of all safety information including vital signs, physical examination, clinical laboratory tests, ECGs, and adverse events.

SUMMARY:
The purpose of this study is to establish single-dose tolerability of inhaled treprostinil sodium in idiopathic pulmonary fibrosis (IPF) patients with pulmonary hypertension, and to explore the acute hemodynamic effects over a range of tolerable doses. The safety and pharmacodynamic information obtained from this study will inform the design and conduct of future studies in inhaled treprostinil sodium in this population.

DETAILED DESCRIPTION:
This is Phase 2, multi-center, open-label, four-cohort study in subjects with pulmonary hypertension (PH) associated with idiopathic pulmonary fibrosis (IPF). Each cohort of four subjects will receive a single dose of inhaled treprostinil sodium. Cohorts will be enrolled sequentially, starting with the lowest dose of 18 mcg. Each cohort escalate by 18 mcg increments, resulting in four cohorts of 18, 36, 54, and 72 mcg doses. Decisions to escalate to the next dose cohort will be based upon the data from the previous completed lower dose cohort of four subjects. Approximately 16 subjects are expected to receive study drug,and approximately four center in the United States with expertise in IPF will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* 35 to 80 years of age
* Male or female
* Diagnosis of IPF

  1. Investigator diagnosis based on history, physical examination, HRCT,and pulmonary function testing
  2. Clinical symptoms of IPF for at least three months prior to Visit 1
  3. High Resolution CT scan showing definite or probable IPF (any time in the past). Bibasilar reticular abnormalities with minimal ground glass opacities on HRCT scan must also be present (at any time in the past)
  4. Surgical lung biopsy showing usual interstitial pneumonia, or transbronchial lung biopsy that was not diagnostic of an alternative condition. For patients younger than 50 years, a surgical lung biopsy is required (at any time in the past)
  5. FVC ≥ 30 % and < 70% of predicted value within three months prior to Visit 1
  6. DLCO ≥ 15% and <70% of predicted value within three months prior to Visit 1.
* Diagnosis of PH

  1. Previously documented radiographic or echocardiographic findings suggestive of pulmonary hypertension
  2. Prior right heart catheterization diagnostic of pre-capillary pulmonary hypertension. [The presence of pre-capillary pulmonary hypertension will be verified by right heart catheterization during Study Visit 3, before enrollment and administration of study drug].
* No changes in concomitant medications prescribed to treat PAH or IPF for 30 days to Visit 1
* Females of childbearing potential may participate only if they are not currently pregnant or lactating and are either one of the following:

  1. Surgically sterile
  2. At least 1 year post-menopausal
  3. Practicing an acceptable method of birth control for at least 30 prior to the Visit 1 with plans to continue this method for the duration of their participation in the study.
* An echocardiogram will be performed at Visit 2. Only those subjects with Visit 2 echocardiographic findings that strongly suggest the presence of pulmonary hypertension, will proceed to Visit 3. Acceptable findings include any of the following:

  1. TR velocity greater than 3.5 m/sec
  2. TR velocity greater than 3.0 m/sec with right ventricular enlargement or dysfunction
* A right heart catheterization will be performed at Visit 3. Only those subjects with Visit 3 right heart catheterization findings that establish the presence of pulmonary hypertension will proceed to enrollment and study drug administration. Acceptable findings must include all of the followings:

  1. mean PA pressure equal or greater than 25 mm HG
  2. pulmonary capillary wedge pressure equal or less than 15 mm Hg
  3. pulmonary vascular resistance greater than 3 mmHg/min

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if ANY of the following criteria apply:

* History of known or suspected pulmonary embolism or deep venous thrombosis
* Clinical evidence of left-sided heart disease
* Presence of atrial fibrillation (determined from 12 lead ECG at Visit 1 or 2)
* Other medical condition or drug exposure known to be associated with pulmonary fibrosis (e.g., rheumatoid arthritis, lupus, scleroderma, etc.) or pulmonary arterial hypertension (e.g., connective tissue disease, congenital heart disease, portal hypertension, HIV infection, drug and toxins, etc.)
* Upper or lower respiratory infection within 30 days prior to Visit 1
* Hospitalization for respiratory illness within 30 days prior to Visit 1
* Diagnosis of any other clinically significant illness that, in the opinion of the investigator, might put the subject at risk of harm from participation in the study or might adversely effect the interpretation of the study data. (e.g., significant liver or kidney disease, etc.)
* History of recurrent symptoms that might, in the opinion of the investigator, adversely effect the interpretation of the study data (e.g., severe headaches, diarrhea, jaw pain, syncope, nausea,vomiting, etc.)
* Current treatment with any medication that is approved by the US FDA to treat pulmonary hypertension (e.g., epoprostenol(Flolan), treprostinil (Remodulin), iloprost (Ventavis), bosentan(Tracleer), ambrisentan (Letairis), sildenafil (Revatio), etc.,), or tadalafil (Cialis)
* Current treatment with an anticoagulant
* A reactive screen for hepatitis B surface antigen, or the hepatitis C antibody, or HIV antibody as tested at Visit 1.
* Use of any inhaled tobacco products or significant history of drug abuse within 90 days prior to Visit 1
* The subject has an echocardiogram performed at Visit 2 that demonstrate findings that are indicative of left ventricular or valvular disease. Findings that will be considered evidence of left ventricular or valvular disease, and therefore exclude the subject from proceeding to Visit 3 are any of the following:

  1. LVEF < 55%
  2. Moderate to Severe mitral regurgitation or aortic regurgitation
  3. Any mitral stenosis or aortic stenosis
  4. Grade 2 or 3 diastolic dysfunction by Doppler
* Use of any investigational drug, or participation in any investigational study within the 30 days prior to Visit 1.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCSD Medical Center m/c7381, La Jolla, California
  - UC Davis Medical Center/Advanced Lung Disease and LungTransplant Program, Sacramento, California
  - University of Michigan, Ann Arbor, Michigan
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UTWS Medical Center Dallas/St. Paul Univ. Hospital, Dallas, Texas
  - Inova Heart and Vascular Institute, Falls Church, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- 18mcg Inhaled Treprostinil Cohort: Patients are to be divided in four cohorts of four patients each. The first cohort will receive a single dose of inhaled Treprostinil (18ug) and each subsequent cohort will receive increasing single doses of 36, 54 and 72ug.
  Each patient will be evaluated on a screening visit (Visit 1) within 28 days prior to dosing, a confirmatory visit (Visit 2) within 14 days prior to dosing, a Baseline/Treatment/Post-Treatment visit( Visit 3) on the dosing day and a Follow-up Period (visit 4) for up to 5 days after dosing.
Period: Overall Study
Arm/Group | 18mcg Inhaled Treprostinil Cohort
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 18mcg Inhaled Treprostinil Cohort
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Inhaled Treprostinil Sodium in Patients With Pulmonary Hypertension Associated With Idiopathic Pulmonary Fibrosis,Reported as Number of Participants With Adverse Events
Description: Safety and Tolerability evaluation include any observed or reported changes in vital signs, ECGs, clinical chemistry ,hematological or urinalysis, and any reported symptoms following a single dose administration on the day of dosing and up to the final visit 3-5 days later. Adverse events will be tabulated by total incidence and by individual patient, and the severity, causality and outcomes will also be documented. Each cohort of 4 patients will be fully evaluated as described before proceeding to the escalation to the next dose.
Time Frame: 3-5 days
Population: Insufficient enrollment, therefore no Participants were analyzed.
Groups:
- 18mcg Inhaled Treprostinil Cohort: Number of participates on a dose of three 6mcg breaths (18mcg total)with Adverse Events
Arm/Group | 18mcg Inhaled Treprostinil Cohort
Number analyzed (Participants) | 0

2. Secondary Outcome: Pharmacokinetic (PK) Parameters After a Single Dose of Inhaled Treprostinil and Acute Hemodynamic Effects.
Description: PK samples will be collected at frequent intervals up to 4 hours following single dosing . Hemodynamic parameters at 4 hours post dosing include heart rate, pulmonary arterial pressure, systemic arterial pressure, right atrial pressure, pulmonary capillary wedge pressure, mixed venous oxygen saturation and cardiac output.
Time Frame: acute
Population: Insufficient enrollment, therefore no participants were analyzed.
Arm/Group | 18mcg Inhaled Treprostinil Cohort
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | 18mcg Inhaled Treprostinil Cohort
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18mcg Inhaled Treprostinil Cohort (N=1)
Headache (General disorders) | 1 (1)
Neck pain at cath site (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was closed on December 31, 2009 and enrolled a total of 1 patient with complete assessment and 4 screened failures. The reason for the closure was lack of enrollment. No data will be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less